CLINICAL TRIAL: NCT03837535
Title: Myocardial Infarction in the Perioperative Setting, a Swedish Multi Center Cohort Study
Brief Title: Myocardial Infarction in the Perioperative Setting
Acronym: MIPS
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Associate Professor, Senior Lecturer, Karolinska University Hospital
Other Study IDs: Karolinska UH_PR
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Myocardial Infarction Postoperative; Myocardial Injury; Intraoperative Complications; Intraoperative Hypotension; Peroperative Complication
MeSH Terms: conditions — Intraoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery: Swedish patients, >18 years undergoing surgery 2007-2014
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Neuro, Lung/thorax, GI, Gynecologic, Urologic, Orthopedic, Vascular surgery

SUMMARY:
Acute myocardial infarction (AMI) is a significant complication following non-cardiac surgery. The investigators sought to evaluate incidence of perioperative AMI, its preoperative and intraoperative risk factors and the outcomes after this complication.

DETAILED DESCRIPTION:
Background:

In Sweden, over 800 000 patients undergo surgery each year. Worldwide, the number of surgical procedures yearly is over 310 million. Surgical care is an essential part of the advancement in treating disease, associated with increased life expectancy and improved quality of life. However, as surgical volume continues to grow, the number of patients who suffer postoperative complications will also increase.

More specifically the project aims to answer the following questions:

1. How common is perioperative acute myocardial infarction following non-cardiac surgery?
2. What are the preoperative and intraoperative risk factors for peroperative AMI?
3. Does perioperative AMI affect mortality and morbidity, Length of stay and days at home?
4. Is the risk of AMI affected by the type of hospital, region or calendar year of surgery?

Orbit - surgical planning system:

The study population was identified from 23 hospitals of all levels (university-, County- and district hospitals) in Sweden, that use the same software program to administer surgical procedures, between 1999 and 2015. The Orbit surgical planning system obligatory includes Swedish identity number, patient demographics, elective or non-elective status, date, type, extent and duration of anesthesia and surgery. Information of the American Society of Anesthesiologists (ASA) physical status classification was often available.

National Patient Register:

To obtain information on discharge dates, covariates and drug exposure, records of surgeries will be linked to the national patient register using the unique Swedish personal identification number assigned to all at birth or at immigration. The national registers have close to complete coverage. The Swedish cause of death registry includes the deaths of all Swedish citizens and residents with a national identity number; it is highly reliable with over 99% of all deaths reported. The Swedish Prescribed Drug Register became operational in July 2005 and contains data on all dispensed prescription of drugs in the Swedish population.

Swedeheart:

To identify all incident cases of myocardial infarctions, the surgical cohort will be linked to Swedeheart, a National Quality Registry containing data on all patients with acute myocardial infarction and all patients undergoing angiographic coronary intervention and heart surgery. The Swedeheart registry was developed in January 1995 and has a present coverage of 95% among incident cases of myocardial infarction treated at a cardiology department.

The National Board of Health and Welfare:

The National Board of Health and Welfare publishes statistics in the areas of health and medical care and social services, including data on acute myocardial infarction. The statistics include all persons aged 20 years and above who have had an acute myocardial infarction reported at the Hospital Discharge Register or the Cause of Death Register. Statistics are presented by year, sex, age and geographical area, information of incidence per 100 000 inhabitants is provided. These data were used to obtain information of expected cases of MI, for standardized incidence ratios (SIR) to be calculated.

Study Participants:

Patients aged 18 years or older undergoing elective or non-elective inpatients surgery between January 1, 2007 and December 31, 2014 were included. Exclusion criteria were surgeries in ambulatory care, cardiac surgery, obstetric- and minor surgical procedures. Patients were also excluded if the surgery was performed prior to 2007 or after 2014, and if a valid surgery code in Orbit - or if a corresponding surgery code in NPR - was lacking.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years), male and female
* Undergoing elective or non-elective inpatient noncardiac surgery

Exclusion Criteria:

* Cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-cardiac surgery between 2007 and 2014 in Swedish Hospitals using the Orbit software surgical planning tool. This software system is used in all parts of Sweden and in all types of hospitals (University, County and District hospitals)
  * University hospitals: Huddinge, KS, Norrlands universitetssjukhus, MAS, USIL, ** County hospitals: NU-sjukvården, Sundsvalls, Södra Älvsborgs, Örnsköldsviks *** District hospitals: Helsingborgs lasarett, Hässleholms, Kristanstads, Kullbergska, Landskrona, Lycksele, Mälarsjukhuset, Nyköping, Sollefteå, Skellefteå Södertälje, Trelleborg, Ystad, Ängelholm, Privat Ortopedisk klinik
Sampling Method: Non-Probability Sample
Enrollment: 400742 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Acute Myocardial Infarction | Within 30days of the index surgery
  AMI, as detected in the postoperative phase in the electronic medical records or in the Swedeheart registry

SECONDARY OUTCOMES:
Mortality | Within 30days of the index surgery and at later predefined time points: 60, 90, 180 and 365 days after the index surgery
  Death, as detected in the postoperative phase in the Swedish cause of death register

OTHER OUTCOMES:
Length of stay (LOS) | LOS within the year after the index surgery
  Time spent in the hospital (number of days)
Days at home alive within 30 days (DAH30) | DAH30 is counted within 30days of the index surgery
  Time spent in the home after the index surgery, takes into account readmissions
Risk of AMI and Mortality by gender, type of surgery, extent- and recency of comorbidity | Within one year of the index surgery
  How above mentioned patient characteristics affect risk of AMI and mortality
Secondary complications | Secondary complications within one year of the index surgery
  AMI vs non-AMI patients and their risk of AKI, pneumonia, stroke, infections, thromboembolic complications
Outcomes (AMI+Mortality+Complications) by hospital, region and year | All outcomes within one year of the index surgery
  All outcomes as affected by hospital type, region and by year

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PhD, Principal Investigator — Karolinska University Hospital, Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified cohort data for primary and secondary endpoints will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within a year of study completion
Access Criteria: Data access will be reviewed by an external research committee at the department of perioperative medicine and intensive care at the Karolinska University Hospital